CLINICAL TRIAL: NCT05109104
Title: Clinical Evaluation of the Sun Protection Factor (SPF) of Sunscreen Products According to the FDA Final Rule: Sunscreen Drug Products (2011)
Brief Title: Clinical Study to Evaluate the Sun Protection Factor (SPF) of Three Sunscreen Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 218005
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-10

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes (erythema) assessor is blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CAP UnScented (Experimental): Single topical application: 80 +/- 2 milligrams (mg) (2.0 +/- 0.05 mg per square centimeter [mg/cm^2]) of CAP UnScented will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: CAP UnScented
- CAP Herbal Mint (Experimental): Single topical application: 80 +/- 2 mg (2.0 +/- 0.05 mg/cm^2) of CAP Herbal Mint will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: CAP Herbal Mint
- CAP Mountain Berry (Experimental): Single topical application: 80 +/- 2 mg (2.0 +/- 0.05 mg/cm^2) of CAP Mountain Berry will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: CAP Mountain Berry
- SPF Standard (Active Comparator): Single topical application: 80 +/- 2 mg (2.0 +/- 0.05 mg/cm^2) of SPF Standard will be applied to the assigned test site using a fingercot. Test material will be evenly spread over the test site using light pressure for 35 +/- 15 seconds.
  Interventions: Drug: SPF Standard Sunscreen

INTERVENTIONS:
Drug: CAP UnScented — Sunscreen lip balm.
  Arms: CAP UnScented
Drug: CAP Herbal Mint — Sunscreen lip balm.
  Arms: CAP Herbal Mint
Drug: CAP Mountain Berry — Sunscreen lip balm.
  Arms: CAP Mountain Berry
Drug: SPF Standard Sunscreen — SPF Standard (7 percent [%] Padimate-O and 3% Oxybenzone)
  Arms: SPF Standard

SUMMARY:
The purpose of this study is to determine the static SPF of three sunscreen products (ChapStick Active Performance [CAP] UnScented, CAP Herbal Mint and CAP Mountain Berry) using the methodology described in the Food and Drug Administration (FDA) Final Rule (2011).

DETAILED DESCRIPTION:
A single-center, randomized, controlled, intra-individual comparison, evaluator-blind, clinical study to determine the SPF of three sunscreen lip balms. Each participant will evaluate the three test products, an SPF standard and no treatment. Study treatments will be randomly assigned to 5 test sites delineated on the skin of the participant's back. Test sites will be exposed to doses of ultraviolet (UV) radiation and erythemal response evaluated 16-24 hours later. Minimal erythema dose (MED) will be determined for protected and unprotected sites and used to determine the SPF value of each test product.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide a signed and dated, legally effective, informed consent document, which indicates they have been informed of all pertinent aspects of the study, before any study procedures are performed.
* Participant must provide relevant details of their medical history and current/recent medications and treatments (self-reported).
* Participant must have completed an annual Health Insurance Portability and Accountability Act (HIPAA) Authorization form.
* Participant must have completed a Photo Release Form.
* Participant must be able to read, write, speak and understand English.
* Participant must be in good general health.
* Participant must have uniform skin color over the test area (skin of the back between the shoulder blades and above the waistline) and an Individual Typology Angle (ITA) value greater than (>)28 degree.
* Participant must have Fitzpatrick Skin Type I, II or III
* Participant must have sufficient area of suitable skin on their back for at least six 40 square centimeter (cm^2) test sites.
* Willing to have body hair clipped by a technician if participant has excessive hair in the test area.
* Participant must have a valid form of personal identification (photo identity [ID], driver's license, passport, permanent resident card, military ID card; forms cannot be expired).
* Male and female participants of child-bearing potential must agree to use a highly effective method of contraception for the duration of the study and for 14 days after their last treatment application. (Note: A participant is considered to be of child-bearing potential if, in the opinion of the principle Investigator [PI], they are biologically capable of having children and sexually active.

Exclusion Criteria:

* Participant with a scheduled or planned Covid-19 vaccination during likely dates of study participation.
* Participant with a history of abnormal response to sunlight/UV radiation.
* Participant with a history of sensitivity to any ingredient of the test material or skin marker pen, or to latex; or any known sensitivities/allergies, including but not limited to cosmetic/toiletry products and topically applied skin treatment products/drugs.
* Participant with any significant dermatological condition, such as atopic dermatitis (eczema), psoriasis, skin cancer, melanoma, active dermal lesions, nevi, blemishes or moles, lupus, diabetes, or connective tissue disease, that would increase the risk associated with participation. (Note: presence of non-dysplastic nevi, blemishes, or moles would be acceptable if, in the opinion of the PI, they will neither jeopardize participant safety or compromise study outcomes. A participant with dysplastic nevi should be disqualified.
* Participant receiving any treatment with medications that would, in the opinion of the PI, confound study outcomes or increase the risk associated with participation, such as systemic or topical corticosteroids, antibiotics, anti- inflammatory drugs, antihistamines, antihypertension medications, or any other photosensitive medications. (Note: The prohibited medication list will be available to site staff for reference during screening).
* Participant who has used topical or systemic steroids, antihistamines, antibiotics or anti-inflammatory medications within 7 days of Study Day 1 which, in the opinion of the PI, could interfere with study outcomes.
* Participant who has used/applied any personal care products (for example, lotions, sunscreens, sunless tanners) and/or topical medications in/on the test area within 24 hours (hrs) of Study Day 1.
* Participant who is unwilling to cease use of personal care products (for example, lotions, sunscreens, sunless tanners) and/or topical medications in/on the test area for the duration of the study.
* Participant with any known communicable disease(s) (for example, Human Immunodeficiency Virus [HIV], Sexually Transmitted Diseases [STD's], Hepatitis B, Hepatitis C, and so on).
* Participant with skeletal protrusions and/or extreme areas of curvature in the test area.
* Participant with a medical treatment/vaccination (other than the Covid-19 vaccination) planned during the study, which would make them ineligible, place them at undue risk, or confound the outcome of the study, per the discretion of the PI.
* Participant who has undergone any surgical procedure in the last 12 months.
* Participant who has undergone chemical or physical treatment procedures in the test area within the last 12 months.
* Planned hospitalization during the study.
* Participant who exceeds a weight limit of 300 pounds due to equipment limitations.
* Participant with any condition that might confound the study results, increase the risk associated with participation, or interfere with study participation.
* Female participant who is pregnant, planning to become pregnant during the study, or breastfeeding (self-reported).
* Participant with any visible sunburn or suntan in test area.
* Participant with visible sun damage, scarring or tattoos in the test area that would interfere with study participation.
* Participant with any sun exposure and/or use of an artificial tanning lamp on the test area within 2 months of Study Day 1.
* Participant who is unwilling to avoid sun exposure and/or cease use of an artificial tanning lamp on the test area for the duration of the study.
* Participant who has participated in any clinical study involving UV exposure within the last 2 months, or any other type of clinical study within the last 1 month.
* Participant who is an employee/contractor or immediate family member of the PI, study site or Sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoint and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United States.
Pre-assignment Details: Study participants were randomly assigned to receive a single topical application of each 4 study treatments (ChapStick Active Performance [CAP] UnScented; CAP Herbal Mint; CAP Mountain Berry and SPF Standard) + 1 untreated site used to determine repeat unprotected Minimal Erythema Dose [MEDuR].
Units Other Than Participants: test sites on back
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of each 4 study treatments (CAP UnScented; CAP Herbal Mint; CAP Mountain Berry and SPF Standard) + 1 untreated site. Each product/untreated test site was delineated on a site on the participants back. Around 80 +/- 2 milligrams (mg) product was applied to each 40 square centimeter (cm^2) test site (2.00 +/- 0.05 mg/cm^2). Test sites received a progressive sequence of timed ultraviolet (UV) radiation exposures and were evaluated for erythema immediately after irradiation and 16-24 hours later. A total of 13 participants were enrolled; 11 received CAP UnScented (11 test sites, of which 1 became invalid); 11 received CAP Herbal Mint (11 test sites, of which 1 became invalid); 13 received CAP Mountain Berry (13 test sites, of which 2 became invalid); 13 received SPF Standard (13 test sites); and 13 participants with 13 untreated test sites (of which 1 became invalid).
Period: Overall Study
Arm/Group | All Study Participants
Started | 13; 61 test sites on back
CAP UnScented | 11; 10 test sites on back
CAP Herbal Mint | 11; 10 test sites on back
CAP Mountain Berry | 13; 11 test sites on back
SPF Standard | 13; 13 test sites on back
Untreated | 13; 12 test sites on back
Completed | 13; 56 test sites on back
Not Completed | 0; 5 test sites on back

BASELINE CHARACTERISTICS:
Population: Safety population: all randomized participants who received at least one dose of a study treatment.
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of each 4 study treatments (CAP UnScented; CAP Herbal Mint; CAP Mountain Berry and SPF Standard) + 1 untreated site. Each product/untreated test site was delineated on a site on the participants back. Around 80 +/- 2 mg product was applied to each 40 cm^2 test site (2.00 +/- 0.05 mg/cm^2). Test sites received a progressive sequence of timed UV radiation exposures and were evaluated for erythema immediately after irradiation and 16-24 hours later. A total of 13 participants were enrolled; 11 received CAP UnScented (11 test sites, of which 1 became invalid); 11 received CAP Herbal Mint (11 test sites, of which 1 became invalid); 13 received CAP Mountain Berry (13 test sites, of which 2 became invalid); 13 received SPF Standard (13 test sites); and 13 participants with 13 untreated test sites (of which 1 became invalid).
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Arithmetic Mean SPF Values
Description: SPF values for each test product and the SPF standard were first calculated for each individual participant:SPFi = MEDp/MEDuR (p=protected [treated] site; u=unprotected [untreated] site). The arithmetic mean SPF, standard deviation (SD) and standard error (SE) were then calculated separately for each test product and the SPF standard from valid SPFi data: SPF = (ΣSPFi)/n; SD = √[(ΣSPFi^2) - ((ΣSPFi)^2/n) /(n-1))]; SE = SD/√n (n = number participants providing valid test results). For SPF determination to be considered valid, in compliance with FDA Final Rule 2011, the mean SPF value of the SPF standard should fall within the SD range of the expected SPF (i.e.,16.3 ± 3.43 or 12.87 to 19.73). The MED is the lowest dose of UV radiation that produces the first perceptible erythema with clearly defined borders (covering more than 50% of the exposure site), 16 to 24 hours (hrs) after UV exposure administration.
Time Frame: From 16 to 24 hours post UV exposure
Population: Analysis Population: all randomized participants who received study treatment and provided valid results. Only those participants who have valid sites were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: test sites on back
Groups:
- CAP UnScented: All participants with valid data for CAP UnScented.
- SPF Standard (CAP UnScented Dataset): All participants with valid data for SPF Standard (CAP UnScented dataset).
- CAP Herbal Mint: All participants with valid data for CAP Herbal Mint.
- SPF Standard (CAP Herbal Mint Dataset): All participants with valid data for SPF Standard (CAP Herbal Mint dataset).
- CAP Mountain Berry: All participants with valid data for CAP Mountain Berry.
- SPF Standard (CAP Mountain Berry Dataset): All participants with valid data for SPF Standard (CAP Mountain Berry dataset).
Arm/Group | CAP UnScented | SPF Standard (CAP UnScented Dataset) | CAP Herbal Mint | SPF Standard (CAP Herbal Mint Dataset) | CAP Mountain Berry | SPF Standard (CAP Mountain Berry Dataset)
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 13 | 13
Number analyzed (test sites on back) | 10 | 10 | 10 | 10 | 11 | 11
Ratio | 29.2 (5.71) | 16.4 (2.27) | 28.2 (4.67) | 16.4 (2.27) | 30.2 (4.05) | 16.4 (2.07)
Statistical Analysis 1: Comparison: CAP UnScented; Test type: Other — The t value from the '2-sided' Student-t distribution table corresponding to the upper 5% point with n-1 degrees of freedom was obtained and the labeled SPF value was determined as the largest whole number less than the following calculation: Labeled SPF = Mean SPF - (t*SE); Labeled SPF = 25
Statistical Analysis 2: Comparison: CAP Herbal Mint; Test type: Other — [test comment as in outcome 1, analysis 1]; Labeled SPF = 25
Statistical Analysis 3: Comparison: CAP Mountain Berry vs SPF Standard (CAP Mountain Berry Dataset); Test type: Other — [test comment as in outcome 1, analysis 1]; Labeled SPF = 27

ADVERSE EVENTS:
Time Frame: From screening until 14 days after last dose administration of trial product (Up to 16 days)
Description: AEs, and therefore all serious adverse events (SAEs), were to be collected from immediately after a participant provided written consent to participate in the trial until 14 days after the last administration of study treatment (or the last study procedure). All SAEs were to be reported within 24 hours of detection. Localized erythema caused by exposure of the skin to UV radiation is expected and was not reported as an adverse event.
Arm/Group | CAP UnScented | SPF Standard (CAP UnScented Dataset) | CAP Herbal Mint | SPF Standard (CAP Herbal Mint Dataset) | CAP Mountain Berry | SPF Standard (CAP Mountain Berry Dataset)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT05109104/Prot_SAP_000.pdf